CLINICAL TRIAL: NCT01550848
Title: A Phase II Study of Abraxane Combined With Gemcitabine in the Patients With Metastatic Breast Cancer
Brief Title: A Phase II Study of Abraxane Gemcitabine Combination in Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xichun Hu, Principal Investigator, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Fudan BR2011-07
Record Dates: First submitted 2012-02-27; First posted 2012-03-12 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Albumin-Bound Paclitaxel; Gemcitabine; Antineoplastic Combined Chemotherapy Protocols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Abraxane and Gemcitabine (Experimental): Abraxane and Gemcitabine
  Interventions: Drug: Abraxane and Gemcitabine

INTERVENTIONS:
Drug: Abraxane and Gemcitabine — ABX (Abraxane) 125 mg/m2，intravenous infusion，30min，day 1, 8, 15
  GEM (Gemcitabine) 800 mg/m2，intravenous infusion，30min，day 1, 8, 15
  Other Names: Combined Chemotherapy

SUMMARY:
The purpose of this study is to evaluate the efficacy and toxicity of Abraxane combined with Gemcitabine in the patients with metastatic breast cancer.

DETAILED DESCRIPTION:
This study is to investigate the efficacy and toxicity of Abraxane combined with Gemcitabine in the patients with metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female between 18 and 70 years old;
* Patients with histologic proved metastatic breast cancer, unsuitable to be treated with surgery;
* ECOG (Eastern Cooperative Oncology Group) 0~1;
* Normal functions with heart, liver,renal and bone marrow:WBC≥3.5×109/L；Hb≥90 g/L；plt≥100×109/L;
* Got ICF (Informed Consent Form) before enrollment;
* Life expectancy more than 12 weeks

Exclusion Criteria:

* Pregnant or breast-feeding women or positive serum pregnancy test;
* Uncontrolled brain metastases. Patients with brain metastases must be locally treated and the disease must be stable for at least one month at the time of enrolling;
* Participation in any investigational drug study within 4 weeks preceding treatment start;
* Concurrent other malignancy at other sites or previous other cancer within the last 5 years, with the exception of adequately treated in situ carcinoma of cervix uteri or basal or squamous cell carcinoma of the skin or a contralateral breast cancer;
* Serious uncontrolled intercurrent infections;
* Poor compliance

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-07 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
overall response rate | 8 weeks

SECONDARY OUTCOMES:
number of adverse events | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Xichun Hu, MD;PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, China

REFERENCES:
- [Derived] Li Y, Zhao Y, Gong C, Xie Y, Hu X, Zhang J, Wang L, Zhang S, Cao J, Tao Z, Wang B. Cisplatin shows greater efficacy than gemcitabine when combined with nab-paclitaxel in metastatic triple-negative breast cancer. Sci Rep. 2019 Mar 5;9(1):3563. doi: 10.1038/s41598-019-39314-y. PMID 30837503
- [Derived] Zhao Y, Lv F, Chen S, Wang Z, Zhang J, Zhang S, Cao J, Wang L, Cao E, Wang B, Hu X. Caveolin-1 expression predicts efficacy of weekly nab-paclitaxel plus gemcitabine for metastatic breast cancer in the phase II clinical trial. BMC Cancer. 2018 Oct 22;18(1):1019. doi: 10.1186/s12885-018-4936-y. PMID 30348118